CLINICAL TRIAL: NCT03694938
Title: Dépistage Des métastases cérébrales Par IRM Chez Les Patients Avec un adénocarcinome Colorectal métastatique
Brief Title: Detection of Brain Metastasis by MRI in Metastatic Colorectal Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DEMECIA
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colon Cancer
Keywords: Brain metastasis; Magnetic resonance imaging
MeSH Terms: conditions — Colonic Neoplasms; Brain Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magnetic resonance imaging (Experimental): Annual MRI during 3 years
  Interventions: Device: Magnetic resonance imaging

INTERVENTIONS:
Device: Magnetic resonance imaging — Annually magnetic resonance imaging

SUMMARY:
The aim of this study is to prospectively determine the incidence of brain metastases in metastatic colorectal cancer patients using systematic annual screening by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven colorectal adenocarcinoma
* Metastases from colorectal cancer diagnosed since less than 6 months
* Indication of an oncologic treatment

Exclusion Criteria:

* Patient with contraindication for MRI
* Diagnosis of cancer other than colorectal cancer in the last three years, except in situ cancers, basal-cell skin cancer or squamous-cell skin cancer, and other cancer with low risk of brain dissemination according to the investigator
* Pregnant or breastfeeding women, women of childbearing potential without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Prospectively determine the incidence of brain metastases in metastatic colorectal cancer patients with annual MRI. | 3 years
  Diagnostic of brain metastases on annual MRI

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - C.H.U. d'Amiens, Amiens
  - Hôpital Privé Jean Mermoz, Lyon
  - C.H.U. de Poitiers, Poitiers
  - C.H.U. de Tours, Tours

IPD SHARING:
Plan to Share IPD: No